CLINICAL TRIAL: NCT05368805
Title: A Phase 1, Open-label, 2-part, 2-period Fixed-sequence Study to Evaluate the Effect of Fruquintinib on the Pharmacokinetics of Dabigatran Etexilate (A P-GP Substrate) and Rosuvastatin (A BCRP Substrate) in Healthy Subjects
Brief Title: Fruquintinib DDI Study With P-gp and BCRP Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-013-00US3
Record Dates: First submitted 2022-04-21; First posted 2022-05-10 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Dabigatran; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): On Day 1, a single oral dose of dabigatran etexilate 150 mg will be given under fasted conditions and serial PK samples will be collected as indicated on the schedule of events. On Day 5, subjects will receive a single oral dose of fruquintinib 5 mg at approximately 1 hour prior to administration of a single oral dose of dabigatran etexilate 150 mg under fasted conditions and serial PK samples will be collected
  Interventions: Drug: Fruquintinib; Drug: Dabigatran Etexilate
- Part B (Experimental): On Day 1, a single oral dose of rosuvastatin 10 mg will be given under fasted conditions and serial PK samples will be collected as indicated on the schedule of events. On Day 5, subjects will receive a single oral dose of rosuvastatin 10 mg with fruquintinib 5 mg under fasted conditions and serial PK samples will be collected
  Interventions: Drug: Fruquintinib; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered as a single oral 5mg dose on the morning of day 5
  Other Names: HMPL-013
Drug: Dabigatran Etexilate — Dabigatran Etexilate will be administered as a single oral dose 150mg on the morning of day 1 and morning of day 5
  Arms: Part A
Drug: Rosuvastatin — Rosuvastatin will be administered as a single oral dose 10mg on the morning of day 1 and the morning of day 5
  Arms: Part B

SUMMARY:
Fruquintinib DDI Study with P-gp and BCRP Substrates

DETAILED DESCRIPTION:
A phase 1, open-label, 2-part, 2-period fixed-sequence study to evaluate the effect of Fruquintinib on the pharmacokinetics of Dabigatran Etexilate (A P-GP substrate) and Rosuvastatin (A BCRP substrate) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.
2. The subject has a body mass index (BMI) >18 and ≤29 kg/m2 at screening.
3. Female subjects must be of non-childbearing potential (eg, postmenopausal [defined as cessation of all menstrual periods for at least 1 year without an alternative medical cause, and confirmed by follicle-stimulating hormone (FSH) test ≥40 IU/L] or surgically sterile by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).
4. Male subjects with partners of childbearing potential must always use a condom and must agree in addition to use a highly effective form(s) of contraception, that results in a low failure rate (<1% per year) when used consistently and correctly, starting during the screening period, continuing throughout the entire study period, and for 90 days after taking the last dose of study drug. Such methods include:

   1. Oral hormonal contraception (combined estrogen/progestogen, or progestogen-only) associated with inhibition of ovulation
   2. Intrauterine device (IUD)
   3. Intrauterine hormone-releasing system (IUS)
   4. Bilateral tubal ligation
   5. Vasectomy
   6. True sexual abstinence in line with the preferred and usual lifestyle of the subject.

   Highly effective contraception should always be combined with an additional barrier method (eg, diaphragm, with a spermicide).
5. The subject must provide written informed consent prior to any study-specific screening procedures.
6. The subject is willing and able to comply with all aspects of the protocol, as determined by the Investigator.

Exclusion Criteria:

1. Clinical laboratory test results from the coagulation panel (international normalized ratio [INR], prothrombin time, and activated partial thromboplastin time) must be within the normal laboratory reference ranges or deemed not clinically significant by the Investigator and Sponsor.
2. The subject has clinically significant renal laboratory findings, including estimated glomerular filtration rate <80 mL/min as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
3. The subject has a known history of any gastrointestinal surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, history of stomach or intestinal surgery or resection). Appendectomy and hernia repair are allowed.
4. The subject had a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
5. The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or at Day -1 check-in (baseline).
6. The subject has systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg.
7. The subject has a clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval >480 msec), or had a family history of prolonged QTc syndrome or sudden death.
8. The subject has a history of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or subject's verbal report and confirmed by cotinine test at check in for each treatment period.
9. The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive urine drug test at screening or at check in for each treatment period.
10. The subject has been diagnosed with acquired immune deficiency syndrome (AIDS) or has performed tests that are positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
11. The subject has participated in a clinical trial of other drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the subject is currently enrolled in another clinical trial.
12. The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
13. The subject has consumed herbal preparations/medications, including, but not limited to, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose.
14. The subject has experienced a weight loss or gain of >10% within 4 weeks prior to the first dose as noted by medical history and weight at screening and check-in.
15. The subject has received blood or blood products within 4 weeks, or donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16 weeks prior to first dose.

    Clinical Study Protocol 2021-013-00US3 Fruquintinib Original Protocol HUTCHMED Limited Page 32 CONFIDENTIAL
16. The subject has used any over-the-counter (OTC) medications or prescription drugs that can affect gastric acid (proton pump inhibitors [PPIs], H2 blockers or locally acting antacids) or that inhibit CYP3A, P-gp, or BCRP in particular, within 2 weeks prior to the first dose.
17. Subject has used CYP3A inducers (including St John's wort) within 30 days before the first dose.
18. The subject is allergic to any of the study drugs (or its excipients) to be given in this study.
19. Female participant is pregnant, lactating, or breastfeeding.
20. Male subject who plans to donate sperm or father a child within 3 months after receiving the study drug.
21. The subject has any condition that would make him or her, in the opinion of the Investigator or Sponsor, unsuitable for the study, or who, in the opinion of the Investigator, is not likely to complete the study for any reason.

One repeat of laboratory assessments may be performed at screening and check in at the discretion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
PK parameter for dabigatran and rosuvastatin: AUC0-t: | Day 1 to Day 13
  area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
PK parameter for dabigatran and rosuvastatin: AUC0-inf: | Day 1 to Day 13
  area under the plasma concentration-time curve from time 0 to infinity (if data permit)
PK parameter for dabigatran and rosuvastatin: Cmax: | Day 1 to Day 13
  maximum observed plasma concentration

SECONDARY OUTCOMES:
Incidence of AEs/SAEs | Day 1 to Day 13
  Any untoward medical occurrence associated with the use of study drug
PK parameter of fruquintinib and metabolite M11: AUC0-t: | Day 1 Day 13
  area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
PK parameters of fruquintinib and metabolite M11: AUC0-inf: | Day 1 to Day 13
  area under the plasma concentration-time curve from time 0 to infinity (if data permit)
PK parameters of fruquintinib and metabolite M11: Cmax: | Day 1 to Day 13
  maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, Austin, Texas, United States